CLINICAL TRIAL: NCT03789409
Title: Intermittent Fasting Following Acute Ischemic Stroke: Prospective, Randomized, Parallel Group, Controlled Trial
Brief Title: Intermittent Fasting Following Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associate Professor, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: chhwang11
Record Dates: First submitted 2018-12-20; First posted 2018-12-28 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Ischemic Stroke; Intermittent Fasting
MeSH Terms: conditions — Ischemic Stroke; Intermittent Fasting

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting (Experimental): Over rehabilitation treatment during and admission (at least 1 week), intermittent fasting (IF) for more than 12 hours (water can be allowed). For subgroup assignment, participants can choose IF1 (eat early in the evening and late in the morning) or Post-IF2 (eat the remaining two meals without breakfast), depending on own their faver.
  Interventions: Dietary Supplement: Intermittent Fasting
- Ad libitium (No Intervention): Participants will be allowed to have hospital meals and all the desired intake without time limit.

INTERVENTIONS:
Dietary Supplement: Intermittent Fasting — The aforementioned intermittent fasting in arm/group descriptions.
  Arms: Intermittent Fasting

SUMMARY:
Despite numerous kinds of evidence on functional health and CNS protection of intermittent fasting after injuries were found in many brain-, and spinal cord-damaged animal models, there has yet to be any clinical study of intermittent fasting after acute ischemic cerebral infarction. The aim of this study is to evaluate the neurological, functional and clinical efficacy of intermittent fasting in patients after acute ischemic stroke.

DETAILED DESCRIPTION:
In order to verify the validity and clinical efficacy of intermittent fasting for neurological and functional effects of ischemic cerebral infarction, the first ischemic stroke (diagnosed within 1 year through brain MRI / CT) patients will be randomly assigned to intermittent fasting group or control group. In both groups, physical therapy, occupational therapy and speech therapy will be provided during 3 hours in total a day. The intermittent fasting group should maintain intermittent fasting for no less than 12 hours or more every day during the rehabilitation period (at least 1 week), and the control group is able to eat all of the hospital meals and all the participants want without any time limit. The efficacy of intermittent fasting is to be verified by performing the electro-physiological tests and functional evaluations before participation, 1st week, 2nd weeks after participation, before discharge, 3 months, and 6 months after the stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was diagnosed first ischemic stroke within preceeding 1 year through brain MRI/CT

Exclusion Criteria:

* Musculo-skeletal disease with limbs malformation or joint contracture
* Weigh more than 135 kg or taller than 195 cm
* Diabetes mellitus
* unstable patient in neurology
* Refusal of participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Surface electromyography | 1 day before the initiation of intervention, and 6 months after the stroke onset
  root mean square and root peak square of compound motor action potential

SECONDARY OUTCOMES:
Change of Korean-modified Barthel index | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Korean version-Modified Barthel Index (minimum of 0 and maximum scores of 100); higher values and a better outcome.

OTHER OUTCOMES:
Change of Mini mental status exam | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Mini mental status exam(minimum of 0 and maximum scores of 30); higher values and a better outcome.
Change of Beck depression inventory | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Beck depression inventory(minimum of 0 and maximum scores of 63); higher values and a worse outcome.
Change of Wecsler aphasia battery | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Wecsler aphasia battery(minimum of 0 and maximum scores of 100); higher values and a better outcome.
Change of Berg balance scale | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Berg balance scale(minimum of 0 and maximum scores of 56); higher values and a better outcome.
Change of Functional Ambulation Category | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Functional Ambulation Category(minimum of 0 and maximum scores of 5); higher values and a better outcome.
Change of Motricity Index | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Motricity Index(minimum of 0 and maximum scores of 99); higher values and a better outcome.
Change of 10m walking test | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  10m walking test
Change of Grasping force (kg) | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Grasping force (kg)
Change of 9-hole pegboard | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  9-hole pegboard
Change of Jebsen Taylor test | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Jebsen-Taylor Hand Function Test
Change of Nottingham sensory scale | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Nottingham sensory scale(minimum of 0 and maximum scores of 20); higher values and a better outcome.
Change of Arm motor Fugl-Mayer scale | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Arm motor Fugl-Mayer scale; wrist & hand/proximal arm(minimum of 0 and maximum scores of 24 and of 34, respectively ); higher values and a better outcome.
Change of Stroke impact scale | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Hand motor, Stroke Impact Scale (minimum of 12 and maximum scores of 60); higher values and a better outcome.
Change of Ashworth scale | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Ashworth scale; elbow, wrist, knee & ankle(minimum of 0 and maximum scores of 4); higher values and a worse outcome.
Change of Knee joint kinesthesia | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  The smallest iso-kinetic angle from which the participants could detect any passive flexion or extension movement of their own knee, using Biodex; (minimum of 0 and maximum scores of 360 degree); higher values and a worse outcome.
Change of Behavioral inatention test | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Behavioral inatention test(minimum of 0 and maximum scores of 146); higher values and a better outcome.
Change of Apraxia screen of Tulia | 1 day before the initiation of intervention and 3rd week after start of intervention, 3 months and 6 months after the stroke onset
  Apraxia screen of (minimum of 0 and maximum scores of 12); higher values and a better outcome.
Change of motor evoked potential | 1 day before the initiation of intervention, and 6 months after the stroke onset
  Amplitude (uV) of motor evoked potential was recorded on abductor pollicis brevis and extentor digitorum brevis following trans-cranial magnetic stimulation for cortico-spinal excitability.
Change of Weight | 1 day before the start of intervention and 1 weeks and 2 weeks after the start of intervention
  Weight (Kg)
Change of Temperature | 1 day before the start of intervention and 1 weeks and 2 weeks after the start of intervention
  temperature (Celsius)
Change of Serum glucose level | 1 day before the start of intervention and 1 weeks and 2 weeks after the start of intervention
  Serum glucose level (mg/ml)
Change of Hypoglycemia-related severity | every day following the start of intervention until 2 weeks of intervention
  Assessment of hypoglycemic symptoms using Likert scale (minimum of 0 and maximum scores of 10); higher values and a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No